CLINICAL TRIAL: NCT05066178
Title: Speech Treatment for Minimally Verbal Children With ASD and CAS
Acronym: TxMVASD+CAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Responsible Party: Principal Investigator, Karen Chenausky, Ph.D., CCC-SLP, Assistant Professor, MGH Institute of Health Professions
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P002598
Record Dates: First submitted 2021-09-16; First posted 2021-10-04 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Developmental Verbal Dyspraxia; Autism Spectrum Disorder
Keywords: childhood apraxia of speech; autism; motor speech disorder; speech development
MeSH Terms: conditions — Apraxias; Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Multiple-baseline single-case design
Masking Description: Outcome assessor will be blinded to participant session
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAS Treatment for MV ASD (Experimental): Participants will receive CAS treatment, modified for minimally verbal children with autism
  Interventions: Behavioral: CAS Treatment for Minimally Verbal Children with Autism

INTERVENTIONS:
Behavioral: CAS Treatment for Minimally Verbal Children with Autism — Treatment involves principles of motor learning embedded in a naturalistic developmental milieu

SUMMARY:
Comorbid Childhood Apraxia of Speech (CAS) may be one factor that limits speech development in some minimally verbal children with autism. CAS is a disorder affecting speech movement planning. This study tests whether CAS-specific treatment, appropriately modified for minimally verbal children with autism, improves their speech.

DETAILED DESCRIPTION:
Although one in four children with autism remain minimally verbal past age five, not all the factors that limit spoken language in these minimally verbal children are known. One powerful contributor may be a motor speech disorder, Childhood Apraxia of Speech (CAS). CAS is an impairment in the ability to plan and sequence for speech, which makes speech inconsistent and imprecise. This project proposes to investigate whether CAS makes the speech of minimally verbal children with autism unintelligible, and then to test whether treating the CAS improves children's speech.

First, a cohort of 20 minimally verbal children with both autism and CAS is identified. The prediction is that the more severe the CAS, the more inconsistent and imprecise a child's speech, and therefore the lower their intelligibility will be. Then, a set of mono- and bisyllabic words is selected that contain the disordered movements that each child shows and use those in treatment.

Treatment will take the form of 15 one-hour sessions where speech practice is embedded in a naturalistic, play-based milieu that is centered on each child's own developmental level. It will involve principles of motor learning (intensive practice of a few words, sometimes all in a row and sometimes mixed up). Different types of cues (touch cues, simultaneous production, etc.) will also be employed to help children say their words correctly, fading back these supports as the child's speech improves. Both of these techniques have been shown to be effective for treating CAS.

Our outcome measures will include both (1) "by-ear" assessments of intelligibility and (2) acoustic and kinematic measurements of children's speech after 15 treatment sessions. The findings will inform clinical practice for minimally verbal children with autism and may lead to the development of novel interventions for this severely affected population.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for Autism Spectrum Disorder
* Able to correctly repeat at least 2 syllables
* Meets criteria for Childhood Apraxia of Speech
* Lives in an environment where child is exposed to English at least 50% of the time

Exclusion Criteria:

* Poorly controlled seizures
* Factors such as blindness or deafness that contribute to minimally verbal status
* Lives in an environment where English is not spoken at least 50% of the time
* Child experiences behavioral challenges that preclude participation in the study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Attempts Correct | 5 weeks
  Number or percent of target items that were produced correctly
Phonemes Correct | 5 weeks
  Number or percent of phonemes (vowels, consonants) in the target items that were produced correctly

SECONDARY OUTCOMES:
Lip aperture movement variability | 5 weeks
  Amount of variability in lip opening area during production of multiple attempts at the same target
Phoneme distinctiveness | 5 weeks
  Acoustic distinctiveness of different phonemes

CONTACTS AND LOCATIONS:
Locations (1):
- MGH Institute of Health Professions, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No